CLINICAL TRIAL: NCT06530199
Title: Simplified Papilla Preservation Flap(SPPF) and Enamel Matrix Derivative(EMD) With or Without Connective Tissue(CTG) Wall for the Treatment of Non Contained Infrabony Defects. A Randomized Controlled Clinical Trail
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02_D012_147502
Record Dates: First submitted 2024-07-19; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Intrabony Periodontal Defect

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Simplified papilla preservation flap with enamel matrix derivative will be performed
  Interventions: Procedure: Enamel matrix derivative
- Test group (Experimental): Simplified papilla preservation flap with connective tissue graft and enamel matrix derivative will be performed
  Interventions: Procedure: Enamel matrix derivative

INTERVENTIONS:
Procedure: Enamel matrix derivative — connective tissue graft and Enamel matrix derivative in the defect area
  Other Names: Connective tissue graft technique

SUMMARY:
Research is to compare and evaluate the clinical and radiographic outcomes of the enamel matrix derivative with or without connective tissue wall graft for noncontained infrabony defects using simplified papilla preservation technique .

DETAILED DESCRIPTION:
Research is to compare and evaluate the clinical and radiographic outcomes of the enamel matrix derivative with or without connective tissue wall graft for noncontained infrabony defects using simplified papilla preservation technique .The objectives is to assess the probing pocket depth reduction, clinical attachment level gain,gingival recession depth and radiographic bone gain. The TEST group will be treated withSIMPLIFIED PAPILLA PRESERVATION flap with connective tissue graft and enamel matrix derivative and the CONTROL group will be treated with SIMPLIFIED APILLA PRESERVATION flap and enamel matrix derivative. The total number of participants included will be 30 (Control-15; Study-15) with a 6 month follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to participate in the study.
* Participants aged ≥18 years to 55 years.
* Presented with non contained infra bony defects.
* Presence of at least 1 non contained infra bony defect(IBD) with a pocket probing depth ≥6mm after reevaluation of the hygienic phase and a depth of IBD ≥3mm as detected on radiographs, with radiographic angulation of ≥37⸰ , and exhibiting a 1 or 2 wall infra bony defect15(assessed by a bone sounding and confirmed intrasurgically)
* Patient's full mouth plaque score and bleeding score <20% at the time of surgical procedure.
* No history of periodontal surgery at the experimental site.

Exclusion Criteria:

* Grade III mobility, endodontically treated teeth.
* Pregnant and lactating females.
* History of tobacco smoking .
* Patients with systemic disease.
* Known allergy or hypersensitivity to EMD.
* Presence of pulpal and peri apical involvement

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
clinical attachment gain | 6 months
  change in attachment level for patient with isolated 2 or 3 wall defect treated with enamel matrix derivative and connective tissue wall graft in 1,3 and 6 months follow up

SECONDARY OUTCOMES:
pocket probing depth | 6 months
  change in pocket probing depth from baseline to 1,3 and 6 months
radiographic bone gain | 6 months
  change in radiographic bone level from baseline to 1,3,6 months
recession reduction | 6 months
  change in recession from baseline to 1,3 and 6 months
plaque index | 6 months
  change in plaque index from baseline to 1,3 and 6 months
gingival index | 6 months
  change in calculus index from baseline to 1,3 and 6 months